CLINICAL TRIAL: NCT01225003
Title: Diffusion Kurtosis Imaging en MR Spectroscopy in Grading and the Characterization of Tumour Infiltration in Gliomas
Brief Title: Advanced MR Techniques in Detection of Tumor Infiltration and Grading in Gliomas
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S52302
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2010-10

CONDITIONS: Gliomas
Keywords: gliomas; magnetic resonance; diffusion kurtosis imaging; MR spectroscopy; grading
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — standard neurosurgical procedure to obtain specimens; standard histopathological examination

SUMMARY:
In this study, we evaluate the role of diffusion kurtosis imaging (DKI) and MR spectroscopy (MRS), two advanced imaging techniques in magnetic resonance (MR) in grading and detection of microscopic infiltrating tumour in gliomas. These parameters are of utmost importance in optimal choice and planning of treatment.

Patients treated with gliomatous brain tumours are included voluntarily. They undergo one imaging session on a 3T MR scanner prior to treatment.

DKI data are quantitively analyzed in order to estimate specific parameters in normal appearing white matter, grey matter, tumor and peritumoral edema. MRS data are analyzed quantitatively and qualitatively with peak integration, ratio calculation and classification algorithms. Histological confirmation is obtained at subsequent surgery.

Information from this study can be of significant importance in avoiding brain biopsies. Furthermore, information on microscopic tumour spread can be used during neurosurgery or in radiotherapy planning. An important advantage of these advanced MR techniques is the non-invasivity and the lack of ionizing radiation, two important issues in this relatively young patient population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of gliomatous brain tumour

Exclusion Criteria:

* younger than 18 years of age
* prior treatment
* history of neurological or neurosurgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with a gliomatuous brain tumor, prior to treatment
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-07

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sunaert, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Uwe Himmelreich, PhD, Principal Investigator — Catholic University Leuven
Locations (1):
- University Hospitals of Leuven, Leuven, Vlaams-Brabant, Belgium